CLINICAL TRIAL: NCT03667859
Title: Vaginal Elasticity Assessment Before and After Brachytherapy/Pelvic Radiation as Measured by Vaginal Tactile Imaging
Brief Title: Vaginal Elasticity Assessment Before and After Brachytherapy/Pelvic Radiation
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0398-18-RMB
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Radiation Injuries
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women undergoing Brachytherapy: Women with either uterine or cervical malignancy treated primarily by brachytherapy.
  Interventions: Diagnostic Test: Vaginal Tactile Imaging
- Women undergoing Pelvic Radiation: Women with either uterine or cervical malignancy treated primarily by pelvic radiation.
  Interventions: Diagnostic Test: Vaginal Tactile Imaging

INTERVENTIONS:
Diagnostic Test: Vaginal Tactile Imaging — Vaginal elasticity measurements using the Vaginal Tactile Imaging system.

SUMMARY:
Female patients with either uterine/cervical malignancies will be evaluated for vaginal elasticity using vaginal tactile imaging both before and after radiation treatment.

DETAILED DESCRIPTION:
Patients will be recruited and sign a consent form. The patients included are patients with either uterine/cervical malignancies. Each participant undergoes radiation treatment either as primary or complementary treatment.

Assessment of vaginal elasticity via vaginal tactile imaging will be performed at 3 different points:

* Before the first treatment session (baseline).
* After the last session of laser treatment.
* 3 months post final treatment. Every patient will serve as her own control. Demographic, gynecologic and obstetric history will be obtained from patients' electronic files.

ELIGIBILITY:
Inclusion Criteria:

* Any woman undergoing either brachytherapy or pelvic radiation treatment as primary or complementary treatment for a cervical/uterine malignancy.

Exclusion Criteria:

* Women that are not in the age range.
* Women with massive vaginal bleeding.
* Women after pelvic exenteration.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with gynecological malignancies.
Study Population: Women undergoing either brachytherapy or pelvic radiation treatment as primary or complementary treatment for a cervical/uterine malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Vaginal elasticity assessment | up to 6 months from enrollment
  Vaginal elasticity as measured by the vaginal tactile imager.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided